CLINICAL TRIAL: NCT03093480
Title: A Non-controlled, Open-Label, Multicenter, Study of Efficacy of rFVIIIFc for Immune Tolerance Induction (ITI) in Severe Hemophilia A Subjects With Inhibitors Undergoing the First ITI Treatment
Brief Title: A Study to Evaluate Efficacy of rFVIIIFc for Immune Tolerance Induction (ITI) in Severe Hemophilia A Participants With Inhibitors Undergoing the First ITI Treatment (verITI-8 Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16473; 2017-000373-36 (EudraCT Number); 997HA402 (Other: Bioverativ Therapeutics Inc.)
Record Dates: First submitted 2017-03-10; First posted 2017-03-28 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia A With Inhibitors
MeSH Terms: interventions — factor VIII-Fc fusion protein; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recombinant coagulation factor VIII Fc (rFVIIIFc) (Experimental): Participants were to receive rFVIIIFc at a dose of 200 international units (IU)/kilogram (kg) as once daily injections or divided on several injections per day at the discretion of the Investigator, starting at baseline visit up to maximum of 48 Weeks in ITI Period. Participants who met the criteria for immune tolerance induction (ITI) success entered the tapering period and received rFVIIIFc at a dose adjusted according to Investigator judgment based on the FVIII activity levels and with the aim of tapering the rFVIIIFc dose to reach a prophylactic dosing regimen within 16 weeks (4 months). Follow-Up was for 32 weeks under an adjusted prophylactic regimen according to Investigator judgment.
  Interventions: Biological: rFVIIIFc

INTERVENTIONS:
Biological: rFVIIIFc — rFVIIIFc 200 IU/kg/day in ITI Period, 50 or 100 IU/kg (adjusted according to Investigator judgement) in tapering Period, and prophylactic regimen in Follow-Up period as powder for injection administered intravenously.
  Other Names: ELOCTATE/ELOCTA; BIIB031; efmoroctocog alfa; antihemophilic factor [recombinant]; Fc fusion protein

SUMMARY:
The primary purpose of this study was to describe the time to tolerization (i.e., ITI success) with rFVIIIFc in participants within a maximum of 48 weeks (12 months) of ITI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability of the participant or his legally authorized representative (e.g., parent or legal guardian) to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local participant privacy regulations
* Male participants of any age diagnosed with severe hemophilia A (as confirmed from the medical record)
* Currently diagnosed with high titer inhibitors (historical peak greater than or equal to (>=) 5 Bethesda units per milliliter (BU/mL), according to medical records)
* Previously treated with any plasma-derived or recombinant conventional or Extended Half-Life FVIII

Exclusion Criteria:

* Other coagulation disorder(s) in addition to hemophilia A
* Previous immune tolerance induction (ITI)
* History of hypersensitivity or anaphylaxis associated with any factor VIII (FVIII) administration
* Planned major surgery scheduled during the study unless deferred until after study completion (minor surgery such as tooth extraction or insertion/replacement of central venous access device is allowed)
* Abnormal renal function (serum creatinine >1.5 milligram per deciliter (mg/dL) or 2 × upper limit of normal (ULN) for participant age based on local laboratory range) as assessed by local laboratory
* Serum alanine aminotransferase or aspartate aminotransferase > 5 × upper limit of normal (ULN) as assessed by local laboratory

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (37):
- United States (12):
  - Center for Inherited Blood Disorders, Orange, California
  - University of Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Dayton Children's Hospital, Dayton, Ohio
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Gulf States Hemophilia and Thrombophilia Center, Houston, Texas
  - Blood Center of Southeast Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Bulgaria (2):
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
- Canada (3):
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- France (5):
  - Hôpital de la Timone, Marseille, Bouches-Du-Rhône
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Hemostase Clinique - Institut Cœur-Poumons (4eme étage aile est), Lille, Nord
  - Hôpital Necker - Enfants Malades, Paris
- Universitaetsklinikum Bonn AoeR, Bonn, North Rhine-Westphalia, Germany
- Italy (3):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Pediatrica Santobono Pausillipon, Napoli
  - Ospedale San Bortolo di Vicenza, Vicenza
- Japan (3):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Nara Medical University Hospital, Kashihara-shi, Nara
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (3):
  - St Thomas' Hospital, London, Greater London
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Royal Hospital for Children, Glasgow, Strathclyde

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Malec L, Van Damme A, Chan AKC, Spasova M, Jain N, Sensinger C, Dumont J, Lethagen S, Carcao M, Peyvandi F. Recombinant factor VIII Fc fusion protein for first-time immune tolerance induction: final results of the verITI-8 study. Blood. 2023 Apr 20;141(16):1982-1989. doi: 10.1182/blood.2022017780. PMID 36735911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 active centers in 7 countries between 08-Dec-2017 to 16-Feb-2021.
Pre-assignment Details: Total 16 participants were screened, enrolled and received drug.
Period: Overall Study
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Started (Immune Tolerance Induction (ITI) Full Analysis Set (ITIFAS): includes all participants who received at least 1 infusion of rFVIIIFc.) | 16
Tapering Period (Tapering Period Full Analysis Set (TPFAS): includes participants entering the tapering phase of the study) | 10
Follow-up Period (Follow-Up Period Full Analysis Set: includes all participants entering the follow-up phase in the study.) | 10
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Based on inclusion criteria, only male participants were included
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Tolerization With rFVIIIFc
Description: Time required for participants to achieve immune tolerance induction (ITI) success where ITI success is defined as achieving all 3 of the following criteria: confirmed negative titers consisting of 2 consecutive negative inhibitor assessments within 2 weeks (less than [<] 0.6 Bethesda units/milliliter [mL] by the Nijmegen-modified Bethesda assay); incremental recovery (IR) greater than or equal to (>=) 66 percent (%) of the expected IR in 2 consecutive assessments; half-life (t½) >= 7 hours.
Time Frame: Up to 48 Weeks
Population: Participants who are in ITI full analysis set (includes all participants receiving at least 1 infusion of rFVIIIFc) and achieved ITI success
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 10
weeks | 11.7 [9.8 to 26.2]

2. Secondary Outcome: Number of Participants With Immune Tolerance Induction (ITI) Success
Description: Number of participants who achieve ITI success where ITI success is defined as achieving all 3 of the following criteria: confirmed negative titers consisting of 2 consecutive negative inhibitor assessments within 2 weeks (<0.6 Bethesda units/mL by the Nijmegen-modified Bethesda assay); incremental recovery (IR) >= 66% of the expected IR at 2 consecutive assessments; half-life (t½) >=7 hours.
Time Frame: Up to 48 Weeks
Population: ITI full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Participants | 10

3. Secondary Outcome: Number of Participants Who Experienced Relapse
Description: Number of Participants with ITI success who reaches the criteria for relapse (defined as confirmed positive inhibitor titer >= 0.6 BU/mL or abnormal recovery after tolerance is achieved, and t½ less than [<] 7 hours) evaluated during the Tapering or Follow-Up Periods
Time Frame: Up to 48 weeks (16 weeks Tapering period and 32 weeks follow-up period)
Population: Tapering Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Annualized Bleeding Rates During ITI Period
Description: A bleeding episode started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. Annualized bleeding rate for a patient during the ITI period is defined as the number of bleeding episodes divided by the length of the ITI period in days* 365.25.
Time Frame: Up to 48 weeks
Population: ITI full analysis set which excludes participants who were observed for less than 90 days during the period
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 13
episodes per participant per year | 6.6 (9.50)

5. Secondary Outcome: Annualized Bleeding Rates After ITI Period
Description: A bleeding episode started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. Annualized bleeding rate for a patient after the ITT period (for tapering and follow-up period) is defined as the number of bleeding episodes divided by the length of the period after the ITI period in days* 365.25.
Time Frame: Up to 48 weeks (16 weeks Tapering period and 32 weeks follow-up period)
Population: Tapering period full analysis set excluding participants who were observed for less than 90 days in the period.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 10
episodes per participant per year
  Tapering period | 1.0 (1.27)
  Follow-up Period | 1.2 (2.91)

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (TESAEs) as a Measure of Safety and Tolerability
Description: An AE is any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition.
Time Frame: Up to 2 Years
Population: ITI full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Participants
  at least one TEAE | 16
  at least one TESAE | 9
  Death | 0
  discontinuation of treatment and/or the study due to an AE | 0

7. Secondary Outcome: Average Number of Days Missed From Work or School Per Month During ITI Period
Description: Average number of days missed from school or work per month for a period (counting in non-missing diary days) is defined as number of the missing school/work days in the period divided by number of days with data entry in the period.
  Number of days per month missed from school or work is reported for those who attend school or have a job.
Time Frame: Up to 48 weeks
Population: Participants of ITI full analysis set and who attend school or have a job
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 3
days | 2.3 (1.21)

8. Secondary Outcome: Average Number of Days Missed From Work or School Per Month After ITI Period
Description: as for outcome 7
Time Frame: Up to 48 weeks (16 weeks Tapering period & 32 weeks Follow-up period)
Population: Participants of Tapering full analysis set and who attended school or have a job
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 1
days | 0 (NA) — Standard deviation cannot be calculated with 1 participant

9. Secondary Outcome: Annualized Number of Hospitalization Days During ITI Period
Description: Annualized number of hospitalization days during a period for a patient is defined as the number of hospitalization days divided by the length of the period in days * 365.25.
Time Frame: Up to 48 weeks
Population: ITI Full analysis set but excluding patients who were observed for less than 90 days in the period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 13
days | 15.4 (32.24)

10. Secondary Outcome: Annualized Number of Hospitalization Days After ITI Period
Description: as for outcome 9
Time Frame: Up to 48 weeks (16 weeks Tapering period & 32 weeks Follow-up period)
Population: Tapering Period Full analysis set but excluding patients who were observed for less than 90 days in the period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 10
days | 2.7 (8.53)

11. Secondary Outcome: Adherence to Treatment Regimen Overall Study Period
Description: Adherence to treatment is based on prescribed daily dose for the overall study period which is defined as the percentage of administered doses versus the prescribed doses to a patient for the entire study duration.
Time Frame: Up to 2 Years
Population: ITI full analysis set
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
percentage of doses | 100.8 (7.76)

12. Secondary Outcome: Annualized rFVIIIFc Consumption for Overall Study Period
Description: Annualized rFVIIIFc consumption for a treatment period is the total nominal rFVIIIFc (IU/kg) / length of period in days * 365.25.
Time Frame: Up to 2 Years
Population: ITI Full analysis set
Measure: Mean (Standard Deviation); unit: international unit (IU)/kilograms (kg)
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
international unit (IU)/kilograms (kg) | 42713.4 (20938.08)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to end of the study (up to 2 years) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent AEs (TEAEs) i.e. defined as AEs that developed, worsened, or became serious on or after the first administration of rFVIIIFc. Analysis performed on ITI full analysis set (ITIFAS).
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 9/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor VIII Fc (rFVIIIFc) (N=16)
Complication associated with device (General disorders) | 1 (1)
Injection site haematoma (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vascular access site infection (Infections and infestations) | 1 (1)
Vascular device infection (Infections and infestations) | 4 (10)
Viral infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (4)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1)
Device breakage (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor VIII Fc (rFVIIIFc) (N=16)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (5)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Eye pruritus (Eye disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (8)
Vomiting (Gastrointestinal disorders) | 3 (3)
Administration site extravasation (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Catheter site extravasation (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (4)
Catheter site swelling (General disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 7 (23)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (3)
Seasonal allergy (Immune system disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (3)
Ear infection (Infections and infestations) | 2 (16)
Gastritis viral (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Myringitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (7)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2)
Tonsillitis (Infections and infestations) | 1 (1)
Vascular device infection (Infections and infestations) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 2 (4)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wrong product administered (Injury, poisoning and procedural complications) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
Serum ferritin decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Device occlusion (Product Issues) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (10)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (9)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4)
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria contact (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03093480/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT03093480/SAP_001.pdf